CLINICAL TRIAL: NCT05295537
Title: Prospective, Randomized, Comparative, Non-inferiority, Multicentre Trial of Quality of Samples Obtained by Percutaneous Liver Biopsy Versus Endoscopic Ultrasound-guided Liver Biopsy
Brief Title: Percutaneous Versus Endoscopic Ultrasound-guided Liver Biopsy (PEREUS)
Acronym: PEREUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, J. Enrique Domínguez-Muñoz, Director of the Department of Gastroenterology, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: USE-01-2021
Record Dates: First submitted 2022-01-16; First posted 2022-03-25 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Liver Diseases
Keywords: Biopsy; Histology; Endoscopic ultrasound; Diagnosis
MeSH Terms: conditions — Liver Diseases; Disease

STUDY DESIGN:
Intervention Model Description: Randomized, parallel assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERCUTANEOUS LIVER BIOPSY (PLB) (Active Comparator): Patients randomized to percutaneous liver biopsy.
  Interventions: Procedure: PERCUTANEOUS LIVER BIOPSY (PLB)
- ENDOSCOPIC ULTRASOUND GUIDED LIVER BIOPSY (EUS - LB) (Experimental): Patients randomized to EUS-guided liver biopsy
  Interventions: Procedure: ENDOSCOPIC ULTRASOUND GUIDED LIVER BIOPSY (EUS-LB)

INTERVENTIONS:
Procedure: PERCUTANEOUS LIVER BIOPSY (PLB) — Percutaneous liver biopsy using a 16 gauge (G) Trucut needle.
  Arms: PERCUTANEOUS LIVER BIOPSY (PLB)
Procedure: ENDOSCOPIC ULTRASOUND GUIDED LIVER BIOPSY (EUS-LB) — EUS-guided liver biopsy using a 19 gauge (G) Franseen core EUS needle
  Arms: ENDOSCOPIC ULTRASOUND GUIDED LIVER BIOPSY (EUS - LB)

SUMMARY:
Although the use of liver biopsy (LB) has decreased with the emerging non-invasive markers and techniques to evaluate liver fibrosis, histopathologic examination of liver tissue is necessary to confirm the type of liver injury. The aim of our study is to compare two methods for obtaining histological material from the liver: the percutaneous liver biopsy (PLB) and the Endoscopic ultrasound (EUS) guided liver biopsy (EUS-LB)

DETAILED DESCRIPTION:
LB remains the gold standard diagnostic test for most of the focal and parenchymal liver diseases. LB has an important diagnostic role in selected parenchymal liver diseases such as autoimmune hepatitis and infiltrative liver disorders, and in some cases, it helps clinicians to elucidate between overlapping diagnoses Traditionally, percutaneous (PLB) or transjugular approaches have been used to acquire liver samples. In recent tears EUS has emerged as an alternative and safe method to obtain liver samples, by puncturing the liver from the gastric or duodenal wall. In fact, EUS-guided LB has been shown equal or superior compared to PLB and transjugular approaches in retrospective series. EUS - LB has shown to produce excellent histological performance based on liver society guidelines requirements for parameters used in assessing histological yield which include the number of complete portal triads (CPT), sample size and total specimen length (TSL) with a low rate of adverse events EUS - LB has several advantages over the traditional liver biopsy methods: it provides simultaneous access to both liver lobes, enables real-time visualization avoiding the puncture of a large vessel and then reducing the rate of complications, it allows to perform a simultaneously endoscopic and endosonography evaluation of the pancreatobiliary system and it could decrease the level of the anxiety of patients (by the use of deep sedation) and then perhaps increasing the satisfaction with the procedure Despite the fact of the high diagnostic yield of EUS-LB in obtaining adequate samples from the liver and the low rate of adverse events reported with this method, there is an almost complete lack of randomized trials comparing EUS - LB with the traditional percutaneous route.

The aim of our study is to compare the quality of samples obtained and the diagnostic efficacy of EUS - LB against PLB in all patients that have an indication for a liver biopsy

ELIGIBILITY:
Patients for whom a liver biopsy have been indicated.

Inclusion Criteria:

* Age over 18 years, any gender
* Understanding and informed consent signed
* Fit for deep sedation

Exclusion Criteria:

* Age below 18 years
* Not signed informed consent
* Contraindication for a deep sedation
* Pregnancy
* Focal liver lesion that requires biopsy visualized by other imaging techniques
* Coagulopathy (INR>1.5 or platelets < 50,000)
* Inability to withdraw anticoagulant or antithrombotic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of tissue samples obtained by EUS-guided liver biopsy compared to percutaneous liver biopsy. | Up to 2 weeks
  The quality of samples is based in the combination of a specimen length >20 mms and more than 10 complete portal triads (both conditions are required).

SECONDARY OUTCOMES:
Diagnostic accuracy of EUS-guided liver biopsy compared to percutaneous liver biopsy. | Up to 2 weeks
  Percentage of samples allowing an adequate histological diagnosis.
Adverse events associated with EUS-guided liver biopsy compared to percutaneous liver biopsy. | At 1 hour, 4 hours, 24 hours, 7 days, and 30 days
  Adverse events evaluated according to the American Society of Gastrointestinal Endoscopy (ASGE) lexicon.
Patient satisfaction after EUS-guided liver biopsy compared to percutaneous liver biopsy. | 24 hours
  Satisfaction survey that includes five points; four are questions scored from 1: bad to 5: excellent; and one is a dichotomic question (Yes/No). Survey will be performed 24 hours after the procedure by phone call.

CONTACTS AND LOCATIONS:
Overall Officials: J. Enrique Dominguez-Muñoz, MD, PhD, Study Director — Hospital Clínico Universitario de Santiago
Locations (1):
- Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No